CLINICAL TRIAL: NCT01818986
Title: Phase II Trial of Sipuleucel-T and Stereotactic Ablative Body Radiation (SABR) for Patients With Metastatic Castrate-resistant Prostate Cancer (mCRPC)
Brief Title: Sipuleucel-T and Stereotactic Ablative Body Radiation (SABR) for Metastatic Castrate-resistant Prostate Cancer (mCRPC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Raquibul Hannan, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 102012-026
Record Dates: First submitted 2013-03-06; First posted 2013-03-27 (Estimated); Results first posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Castrate-resistant Prostate Cancer; mCRPC
MeSH Terms: interventions — sipuleucel-T

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- arm one (Experimental): Sipuleucel-T and Stereotactic Ablative Body Radiation (SABR)
  Interventions: Drug: Sipuleucel-T; Radiation: Stereotactic Ablative Body Radiation

INTERVENTIONS:
Drug: Sipuleucel-T
  Other Names: Provenge
Radiation: Stereotactic Ablative Body Radiation
  Other Names: SABR

SUMMARY:
In this i-SABR (immunotherapy + Stereotactic Ablative Body Radiation) trial, the stereotactic radiation to multiple metastatic sites is delivered not only to eradicate sites of bulky progressive disease, but also to provide antigen presentation and immune stimulation which is expected to act synergistically to the concurrently administered immunotherapy Sipuleucel-T and thereby significantly improve the treatment outcome for metastatic castrate resistant prostate cancer patients (mCRPC). Both Sipuleucel-T and SABR are FDA approved therapeutic cancer treatment

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven prostate cancer
2. Patient must currently be on androgen deprivation or anti-androgen therapy with castrate levels of testosterone (< 50ng/dl). Medical castration should continue until disease progression
3. Radiographic evidence of metastatic disease documented with bone scan or CT scan. Patients with any number of metastatic site are allowed to enroll. However, only up to six sites will be selected for SBRT treatment, at the discretion of the treating radiation oncologist.
4. PSA ≥ 5 ng/ml
5. Asymptomatic or minimally symptomatic patients1. Visual Analog Scale (VAS) ≤ 4;vNo narcotic use in the last 21 days
6. Adequate hematologic, renal, and liver function
7. Previous treatment with surgery, radiation or hormonal therapy is allowed.
8. Performance status ECOG 0 or 1.
9. Life expectancy of at least 6 months
10. Negative serology tests for human immunodeficiency virus (HIV) 1 and 2, human T cell lymphotropic virus (HTLV)-1, Hepatitis B and C.
11. Age ≥ 18 years.
12. Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

1. Subjects must not have had more than two different regiments of chemotherapy previously or any chemotherapy within the past three months.
2. Subjects may not be receiving any other investigational agents for the treatment of prostate cancer.
3. Subjects with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
4. Subjects with malignant pleural effusions and malignant ascites
5. Systemic corticosteroid use within past 28 days. Use of inhaled, intranasal, and topical steroids is acceptable.
6. Systemic immunosuppressive therapy in the past 28 days.
7. Use of any of the following within the past 28 days: Megestrol acetate (Megace®), diethyl stilbestrol (DES), or cyproterone acetate, Ketoconazole, high dose calcitriol [1,25(OH)2VitD] (i.e., > 7.0 μg/week).
8. Inability to tolerate contrast dye for baseline CT imaging.
9. Initiation or discontinuation of biphosphonate use within past 28 days.
10. Subjects with pathologic long-bone fractures
11. Subjects with spinal cord compression
12. Paget's disease of bone.
13. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07-10 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2021-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raquibul Hannan, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sipuleucel-T and SABR (Stereotactic Ablative Body Radiation): Sipuleucel-T (brand name Provenge) IV infusion and Stereotactic Ablative Body Radiation (SABR) dose varying from 21 Gy-33 Gy in 1-3 fractions.
Period: Overall Study
Arm/Group | Sipuleucel-T and SABR (Stereotactic Ablative Body Radiation)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm One: Sipuleucel-T and Stereotactic Ablative Body Radiation (SABR)
  Sipuleucel-T
  Stereotactic Ablative Body Radiation
Arm/Group | Arm One
Number analyzed (Participants) | 20
Age, Customized [Mean (Standard Deviation); unit: years]
  Age at Enrollment | 69 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, not Hispanic | 14
  Black, not Hispanic | 4
  Hispanic | 1
  Asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 20
Baseline performance status [Count of Participants; unit: Participants] — Zubrod Performance Scale will be used:
  0 Fully active, able to carry on all predisease activities without restriction;
  1. Restricted in physically strenuous activity but ambulatory and able to carry work of a light or sedentary nature. For example, light housework, office work;
  2. Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours;
  3. Capable of only limited self-care, confined to bed or chair 50% or more of waking hours;
  4. Completely disabled. Cannot carry on self-care. Totally confined to bed;
  5. Death
  Participants
    0 | 12
    1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: To evaluate the improvement in the time to progression (TTP) of metastatic prostate cancer after the combined treatment with sipuleucel-T and SABR to metastatic sites, as compared to the historically reported data with the treatment of sipuleucel-T alone. Progression will be evaluated in this study using the modified new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) Committee [JNCI 92(3):205-216, 2000] with modifications suggested by PCWG2 [49] recommendations and as used in the Phase III clinical trial by Kantoff et. al.[10]. Changes in only the largest diameter (one-dimensional measurement) of the tumor lesions are used in the RECIST v1.1 criteria as outlined in http://www.recist.com/.
Time Frame: 4 years
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sipuleucel-T and SABR (Stereotactic Ablative Body Radiation)
Number analyzed (Participants) | 20
weeks | 11.2 [6.8 to 14.0]

2. Secondary Outcome: Immune Response
Description: To evaluate the percentage of participants with Immune response at 6 weeks. Immune response will be measured using ELISpot assay (with PA2024). An immune endpoint will be reached by the patient if a >100% increase in immune response is measured by ANY of the assays.
Time Frame: 6 week
Measure: Number; unit: percentage of participants
Arm/Group | Sipuleucel-T and SABR (Stereotactic Ablative Body Radiation)
Number analyzed (Participants) | 16
percentage of participants | 50

3. Secondary Outcome: Overall Survival (OS)
Description: To evaluate the improvement in the overall survival (OS) of mCRPCa patients after the combined treatment with sipuleucel-T and SABR to metastatic sites, as compared to the historically reported data with the treatment of sipuleucel-T alone. Overall survival (OS) was defined as the duration of time from the start of treatment to the time of death from any cause.
Time Frame: 60 months
Measure: Median (95% Confidence Interval); unit: number of weeks
Arm/Group | Sipuleucel-T and SABR (Stereotactic Ablative Body Radiation)
Number analyzed (Participants) | 20
number of weeks | 76.8 [41.6 to 130.8]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: To evaluate the improvement in the progression free survival (PFS) of mCRPCa patients after the combined treatment with sipuleucel-T and SABR to metastatic sites, as compared to the historically reported data with the treatment of sipuleucel-T alone. Progression free survival (PFS) was defined as the length of time from the start of treatment to disease progression or death from any cause.
Time Frame: 4 years
Measure: Median (95% Confidence Interval); unit: number of weeks
Arm/Group | Sipuleucel-T and SABR (Stereotactic Ablative Body Radiation)
Number analyzed (Participants) | 20
number of weeks | 10.4 [6.4 to 13.9]

5. Secondary Outcome: Biochemical Progression Free Survival (bPFS)
Description: To evaluate the improvement in the biochemical progression free survival (bPFS) of mCRPCa patients after the combined treatment with sipuleucel-T and SABR to metastatic sites, as compared to the historically reported data with the treatment of sipuleucel-T alone. Biochemical progression free survival was defined as the time from the beginning of treatment to PSA (prostate-specific antigen) disease progression. Biochemical progression was defined as an increase in PSA of > 2 ng/ml from baseline and an increase of > 25% from the baseline value and confirmed by a second measurement more than three weeks later.
Time Frame: 4 years
Measure: Median (95% Confidence Interval); unit: number of weeks
Arm/Group | Sipuleucel-T and SABR (Stereotactic Ablative Body Radiation)
Number analyzed (Participants) | 20
number of weeks | 12.5 [4.8 to 33.5]

6. Secondary Outcome: Prostate Cancer-specific Survival (PCaSS)
Description: To evaluate the improvement in the prostate cancer-specific survival (PCaSS) of mCRPCa patients after the combined treatment with sipuleucel-T and SABR to metastatic sites, as compared to the historically reported data with the treatment of sipuleucel-T alone. Prostate cancer-specific survival was defined as the percentage of patients who had not died from prostate cancer at the time of analysis
Time Frame: 4 years
Measure: Number; unit: percentage of participants
Arm/Group | Sipuleucel-T and SABR (Stereotactic Ablative Body Radiation)
Number analyzed (Participants) | 20
percentage of participants | 5

7. Secondary Outcome: Adverse Events
Description: To evaluate the adverse events for the first 6 months after completion of radiation therapy associated with Sipuleucel-T when administered in combination with SABR to metastatic sites, as compared to the historically reported data with the treatment of Sipuleucel-T alone. Toxicity will be assessed according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 4.0. Adverse events not specifically defined in the NCI CTCAE will be scored on the Adverse Event log according to the general guidelines provided by the NCI CTCAE and as outlined:
  Grade 1: Mild Grade 2: Moderate Grade 3: Severe or medically significant but not immediately life threatening Grade 4: Life threatening consequences Grade 5: Death related to the adverse event
Time Frame: 60 months
Measure: Number; unit: number of events
Arm/Group | Sipuleucel-T and SABR (Stereotactic Ablative Body Radiation)
Number analyzed (Participants) | 20
number of events
  Grade 1 | 51
  Grade 2 | 8
  Grade 3 | 4

8. Secondary Outcome: Cost Effectiveness and Health-related Quality Adjusted Life
Description: To evaluate the cost effectiveness and health-related quality adjusted life of the combination treatment of SABR and sipuleucel T in patients with mCRPC.
Time Frame: 4 years
Population: This data was not collected per protocol. The objective in question was intended to be an exploratory objective rather than a primary objective. However, due to an error in protocol modification, this change did not occur.
Arm/Group | Sipuleucel-T and SABR (Stereotactic Ablative Body Radiation)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 60 months. Each patient will be assessed for the development of toxicity for 6 months following the completion of radiation therapy and 60 months for overall survival.
Description: Adverse events will be graded by a numerical score according to the defined NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe or medically significant but not immediately life threatening; Grade 4: Life threatening consequences; Grade 5: Death related to the adverse event
Arm/Group | Arm One
All-Cause Mortality (participants affected / at risk) | 19/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm One (N=20)
Alkaline Phosphatase Increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chills (General disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Fatigue (Nervous system disorders) | 11 (11)
Fever (General disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headaches (Nervous system disorders) | 1 (1)
Hot Flashes (Vascular disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Lymphocyte Count Decrease (Investigations) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (6)
Non-Cardiac Chest Pain (General disorders) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Rectal Pain (Gastrointestinal disorders) | 1 (1)
Rectal Urgency (Gastrointestinal disorders) | 1 (1)
Thrombolic Event (Vascular disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Urinary Tract Obstruction (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
White blood cells decreased (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-05): https://cdn.clinicaltrials.gov/large-docs/86/NCT01818986/Prot_SAP_000.pdf